CLINICAL TRIAL: NCT04879056
Title: Instrument Precision Study for Validation of PIPS 5.1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Philips Digital & Computational Pathology (Industry)
Responsible Party: Sponsor
Other Study IDs: 10254
Record Dates: First submitted 2021-01-25; First posted 2021-05-10 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pathology
Keywords: WSI; features

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intra-system: reviewing selected features on images from three iterations of the same scanner.
  Interventions: Diagnostic Test: PIPS 5.1
- inter-system: reviewing selected features on images from three different scanners.
  Interventions: Diagnostic Test: PIPS 5.1

INTERVENTIONS:
Diagnostic Test: PIPS 5.1 — Description: Scanning glass slides on PIPS 5.1. This intervention will be applied in the arm of intra-system and the arm of inter-system.

SUMMARY:
This study is designed to evaluate the instrument precision of the device for its proposed intended use in sub-studies: intra-system and inter-system. The precision within a system will be evaluated on three systems by three pathologists at one site. Specific features will be selected on glass slides, which will then be scanned. On the whole slide images field of views will be created including the features. In the reading phase three pathologists will read the field of views and record which features they observe.

DETAILED DESCRIPTION:
This study is designed to evaluate the instrument precision of the device for its proposed intended use in sub-studies: intra-system and inter-system. Each sub-study will have three phases: enrollment, preparation and reading.

Per sub-study the precision of the device will be based on three reading pathologists' assessments and identification of specific clinically relevant histopathologic "features" that are encountered in formalin-fixed, paraffin-embedded (FFPE) hematoxylin and eosin (H&E) slides. Examples of these features are eosinophils, plasma cells, goblet cells, foreign body giant cells, etc. Three magnifications are used in this study: 10x, 20x and 40x. These magnifications represent the magnifications typically used in routine clinical practice. There will be seven different study features per magnification. In total twenty-one features will be selected, with each feature selected from at least three different organs, to ensure that multiple tissue types are investigated.

Precision will be assessed in sub-studies: intra-system and inter-system.

1. In the intra-system study the precision within a system will be evaluated on three systems by three pathologists at one site;
2. In the inter-system study the precision between systems will be evaluated on three systems by three pathologists at one site;

Enrollment:

The enrollment process (case selection, slide selection, feature selection, and field of view (FOV) selection) will be performed by an enrollment pathologist (EP), a validating enrollment pathologist (VEP) and a study technician.

Cases will be selected from the laboratory information system (LIS) by the EP. For each pre-specified study feature and organ, consecutive cases will be selected per feature. From these cases, slides will be selected containing the pre-specified study feature(s) for which the EP is searching at that moment. The study feature(s) on the chosen slide is/are then called the "selected feature(s)". The VEP confirms if the selected feature(s) is/are present on the glass slide. The validated slides are scanned by a study technician for enrollment. The EP reviews the whole slide image (WSI) of the slide and defines an area (bookmark) containing the selected feature(s) at the appropriate magnification. The sponsor will create a static full resolution extraction image of the bookmark, which will then be defined as the FOV. The VEP confirms if the feature(s) is/are present on the FOV. Note that the precise flow may be adapted according site preference with the pre-requisite that all slides and FOVs are selected and validated before enrolment. After confirmation, the FOV is considered enrolled.

Scanning and reading:

After enrollment the slides are scanned by the study technician for the reading sessions. The sponsor extracts the FOV(s) from each image, identical to the enrollment FOV. Scanning and reading will be different per sub-study, see below.

The reading pathologists in this study will be blinded to certain details in the protocol e.g. the study features.

The reading pathologist will review the FOV as a snapshot with no panning or zooming capabilities. The reading pathologist will assess the presence of each of the features on a feature checklist appropriate for that particular magnification.

Scanning and reading intra-system study:

The study slide set will be equally (n=133 slides per system) and randomly divided over three systems at one site. On each system the slides are scanned three times with at least six hours of system downtime (ensuring full cool down) between scanning iterations.

Three separate reading sessions will be performed by each of three reading pathologists, with a washout period of at least two weeks between individual sessions.

Each reading pathologist will read all study FOVs from all three iterations and all three systems in a randomized way.

Scanning and reading inter-system study:

The complete study slide set (n=399) will be scanned once on each of the three systems at one site. Three separate reading sessions will be performed by each of the three pathologists with a washout period of at least two weeks between individual sessions. Each reading pathologist will read all study FOVs in a randomized way.

ELIGIBILITY:
Inclusion Criteria:

* Left-over specimens from subjects who already received their diagnosis and have received their treatment in accordance with the standard of care
* H&E glass coverslipped slides with human tissue obtained via surgical pathology
* Selected slides fulfill the quality checks according to the IfU
* Selected slides must be at least one year since accessioning
* Selected slides and FOVs must contain a study feature that is:

  * In it's natural environment (on slide and FOV)
  * Not equivocal (on slide and FOV)-

Exclusion Criteria:

* Selected slides contain indelible markings
* Selected slides contain damaged tissue
* More than one slide was selected for a patient (only one slide may be enrolled per patient).

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study features are selected on glass slides from consecutive cases from the laboratory information system.
Sampling Method: Probability Sample
Enrollment: 399 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of features | 1 day
  Each reading pathologist will record the presence of listed features on the checklist. The results will be used for deriving an agreement rate between repeated readings from the same reading pathologist over all enrolled (i.e. selected and validated) features.

CONTACTS AND LOCATIONS:
Overall Officials: Mischa Nelis, MsC, Study Director — Philips Digital & Computational Pathology
Locations (1):
- Capital Choice Pathology Laboratory, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No